CLINICAL TRIAL: NCT03102372
Title: Preservation of Fat Free Mass During Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Orkla Health (Unknown); Toyota-Fonden (Other); Tømmerhandler Vilhelm Bangs Fond (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Section of Sport Science, AU
Record Dates: First submitted 2017-03-10; First posted 2017-04-05 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Muscle Loss
Keywords: FFM; VLCD; exercise; Protein; Obesity
MeSH Terms: conditions — Muscular Atrophy; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized single blinded, controlled intervention trial
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein group (Experimental): 4 weeks of a Very Low Calorie Diet (VLCD) + walking program. Whey protein supplementation 0.4g/kg before sleep.
  Interventions: Dietary Supplement: Whey protein supplementation; Other: walking program; Other: Very Low Calorie Diet
- Placebo group (Placebo Comparator): 4 weeks of a Very Low Calorie Diet (VLCD) + walking program
  Interventions: Other: walking program; Other: Very Low Calorie Diet

INTERVENTIONS:
Dietary Supplement: Whey protein supplementation
  Arms: Protein group
Other: walking program
Other: Very Low Calorie Diet

SUMMARY:
In this study, we aimed to examine the effect of whey protein supplementation given before night sleep on Fat Free Mass (FFM) preservation during a 4 wk period on Very Low Caloric Diet (VLCD).

Half of the participants underwent a 4 week VLCD and walking program, while the other half underwent a 4 week VLCD, walking program and had an additional protein supplement before each night sleep.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (kg/m^2) > 28
* Age between 18 and 55 years

Exclusion Criteria:

* Participation in regular resistance-, aerobic- or anaerobic training (>1 h/wk within the last 3 month before intervention start)
* Diabetes Physical disabilities that would hinder completion of the walking program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Fat Free Mass | Change from baseline to after the 4 week intervention period
  Dual energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Nitrogen balance | Change in nitrogen content from baseline to day 7 and 28 of the intervention period
  Three 24 hours urin samples
Oral glucose tolerance test | Change from baseline to after the 4 week intervention period
  OGTT
Fitness level | Change from baseline to after the 4 week intervention period
  Bike test
Blood pressure | Change from baseline to after the 4 week intervention period
  Blood pressure at rest
Fat mass | Change from baseline to after the 4 week intervention period
  DXA
waist circumference | Change from baseline to after the 4 week intervention period
  waist circumference
Performance test | Change from baseline to after the 4 week intervention period
  Intermittent running test (YY1R1C)

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, Lector, Principal Investigator — Aarhus University, Department for Public Health, Section for Sport Science

IPD SHARING:
Plan to Share IPD: No